CLINICAL TRIAL: NCT01622972
Title: Mode of Action of Moviprep:Impact on Distribution of Intestinal Fluid and Colonic Microbiota
Brief Title: Mode of Action of Moviprep
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: Norgine (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 10050; 2010-021879-85 (EudraCT Number)
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Last update posted 2014-04-14 (Estimated); Status verified 2014-04

CONDITIONS: Functional Constipation; Irritable Bowel Syndrome Characterized by Constipation
MeSH Terms: interventions — polyethylene glycol 3350; MoviPrep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): Healthy volunteers in Group 1: To give sachet's A and B made up to 1 litre with tap water once on day 1 and once on day 2
  Interventions: Drug: Polyethyleneglycol
- Group 2 (Experimental): Healthy volunteers in group 2: To give 2x sachet's A and B made up to 2 litres with tap water on day 1.
  Interventions: Drug: Polyethyleneglycol
- Group 3 (Experimental): Patients with functional constipation and irritable bowel syndrome characterized by constipation: To give sachet's A and B made up to 1 litre with tap water once on day 1
  Interventions: Drug: Polyethyleneglycol

INTERVENTIONS:
Drug: Polyethyleneglycol — Group 1 sachet's A and B made up to 1 litre with tap water once on day 1 and once on day 2. Group 2 2x sachet's A and B made up to 2 litres with tap water on day 1. Group 3 sachet's A and B made up to 1 litre with tap water once on day 1.
  Other Names: Macrogol 3350; Moviprep

SUMMARY:
The University of Nottingham have been developing new, non-invasive magnetic resonance imaging (MRI) techniques to image the bowel. Building on those studies the investigators want to study, in healthy volunteers, the effects of purging on the colon. The investigators plan two studies using their novel MRI techniques in healthy volunteers to demonstrate how doses of a preparation designed to clean the bowel alters small and large bowel water content and transit. The investigators will also define the changes induced in colonic microbiota and how these are linked to changes in transit and the structure of colonic contents. This experimental model is comparable to an episode of acute diarrhea, therefore this study will also improve their understanding of the effects of diarrhea on bowel physiology.

Following from the above study, the investigators would like to extend this study on patients who have functional constipation and previously have not responded to conventional laxatives.

DETAILED DESCRIPTION:
Routine examinations of the colon including colonoscopy and barium enema widely carried out in clinical practice require evacuation of colonic contents. This is most conveniently carried out using osmotic laxatives the most widely used preparation being based on polyethylene glycol such as Moviprep. When fully made up as 1 litre of Moviprep , it provides 100 grams of polyethlene glycol '3350' with a measured osmolarity of around 530 mosmol/l. Being nonnutrient, this would be expected to rapidly leave the stomach and generate a substantial inflow of fluid in the upper small intestine as water flows down the osmotic gradient markedly increasing the small intestinal water content compared with fasting.

Previous MRI studies using a Mannitol solution of 300 mosmols/l resulted in a small bowel secretion of fluid increasing total small bowel water to nearly 400 mls after a 300 ml meal. The investigators would anticipate a much larger increase after the hypertonic Moviprep. The flush of small bowel fluid induced by mannitol produces a radical change in the heterogeneous structure of the ascending colon as shown in our recent MRI images of the colon before and after mannitol.

Contrary to expectation colonic contents are far from homogenous with a spatially organised bacterial flora which others have described at a microscopic level which the investigators are just beginning to demonstrate using their novel MRI techniques. The colon should be regarded as a complex bioreactor which is spatially highly organised with a mucous layer overlying the enterocytes, the outer layer of mucus containing a germinal layer with bacteria which reseed the bioreactor when it is purged. The rate of recovery after purgation with polyethylene glycol is said to be normally rapid as the intact germinal layer rapidly recolonises but slower in certain patient groups though data is very limited as yet. The anecdotal yet persuasive patient accounts of improvement in bowel function after colonic lavage suggest that the reconstituted microbiota may be different, though this has yet to be studied using modern techniques.

Until recently the investigators have had no way of noninvasive imaging this complex structure but recent developments of high resolution MRI in Nottingham show that this is now feasible. Pilot data demonstrates that purging removes the heterogeneous three dimensional structure leaving homogeneous fluid contents with an intense proton signal. Just how this impacts on the colonic microbiota is as yet unknown as there have been no studies to date combining these novel approaches with new techniques now available for assessing the microbiota.

Early culture-based assessments identify only a minority of all the faecal organisms present and it is only in the last decade that methods based on assessment of microbial DNA have evolved to make it possible to describe the full complexity of the faecal microbiota. PCR of the highly conserved 16s ribosomal RNA gene shows the microbiota of individuals to be highly complex and individualised. Similarity indices show similarities of around two thirds over a 7 week period in healthy controls while those developing acute diarrhoea due to radiation enteritis show a marked reduction to just 26%. Similarly, HITChip analysis showed that subjects with IBS had an unstable microbiota that was stabilised following a probiotic intervention trial that improved the IBS symptom score. These techniques have yet to be applied to subjects undergoing bowel purgation. Moreover, there are novel approaches to identify the viability of the microbiota such as the use of specific probes that allow discrimination between intact, damaged and dead cells in fecal samples.

ELIGIBILITY:
Inclusion Criteria Group 1 and 2:

* Male or female healthy volunteers who are 18-65 years
* BMI 18-28 kg/m2
* Able to give voluntary written informed consent to participate in the study
* Able to understand the requirements of the study, including anonymous publication, and agree to co-operate with the study procedures

Inclusion Criteria Group 3:

* Male or female who are 18-65 years
* BMI 18-30 kg/m2
* Able to give voluntary written informed consent to participate in the study
* Able to understand the requirements of the study, including anonymous publication, and agree to co-operate with the study procedures
* Patient diagnosed with constipation predominant irritable bowel syndrome who failed to respond to at least 1 laxative treatment in the past
* Patient diagnosed with functional constipation who failed to respond to 1-2 sachets of Movicol per day

Exclusion Criteria for group 1 and 2:

* Any history of serious acute or chronic illness especially gastrointestinal
* Diabetes Mellitus
* Pregnancy or breast feeding
* Smoking
* Unsuitable for MRI scanning (i.e. have metal implants or a pace maker)
* Regular use of medication interfering with gastrointestinal function including opiates or constipating drugs
* Subjects using the oral contraceptive pill will be excluded if not prepared to use an alternative barrier method of contraception for the duration of the menstrual cycle following dosing with Moviprep
* Substance abuse
* Have taken part in another clinical study within the previous 3 months
* Previous gastrointestinal surgery of any kind apart from appendicectomy

Exclusion criteria for group 3:

* Any history of serious acute or chronic illness especially gastrointestinal
* Diabetes Mellitus
* Pregnancy or breast feeding
* Unsuitable for MRI scanning (i.e. have metal implants or a pace maker)
* Regular use of medication interfering with gastrointestinal function including opiates or constipating drugs
* Subjects using the oral contraceptive pill will be excluded if not prepared to use an alternative barrier method of contraception for the duration of the menstrual cycle following dosing with Moviprep
* Substance abuse
* Have taken part in another clinical study within the previous 3 months
* Previous gastrointestinal surgery of any kind apart from appendicectomy/cholecystectomy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2011-09; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Effect of 1 or 2 litre of Moviprep on area under curve (AUC) small bowel water content 0-6 hours on healthy volunteers | up to 24 hours
  Healthy Volunteers
To assess area under curve of small bowel water content following 1litre of Moviprep on patients with constipation | up to 6 hours
  Patients with constipation

SECONDARY OUTCOMES:
Effect of 2 different dosing regimens of Moviprep on cleansing of the colon as assessed from colonic contents on the last scan at the end of purgation | up to 24 hours
  Healthy volunteers
Effect of 2 different dosing regimens of Moviprep on the time course of the intestinal water content | 6 weeks
  Healthy volunteers
Effect of 2 different dosing regimens of Moviprep on the time course of the ascending colon total chyme volume | 6 weeks
  healthy volunteers
Effect of 2 different dosing regimens of Moviprep on the time course of the Colonic motility index 'cine' MRI movies | 6 weeks
  Healthy volunteers
Effect of 2 different dosing regimens of Moviprep on the time course of the transit assessment from mean position of marker capsules | 6 weeks
  Healthy volunteers
Comparison of single dose versus split dose on above MRI parameters | 6 weeks
  healthy volunteers
Rate of recovery of normal colonic microbiota over days 2-28 assessed by bacterial DNA data (HITChip) and SCFA concentration | 6 weeks
  healthy volunteers
Correlation between microbiota, SCFA and colonic MRI parameters | 6 weeks
  Healthy volunteers
Ascending colon total chime volume | up to 6 hours
  Patient with constipation
Colonic motility index 'cine; MRI movies | up to 6 hours
  Patients with constipation
C) Comparison of the cross sectional area of the ascending colon with the cross sectional area of the transverse and descending colon | up to 6 hours
  Patients with constipation
Transit assessment from mean position of marker capsules at 24 hours | 24 hours
  Patients with constipation

CONTACTS AND LOCATIONS:
Overall Officials: Robin Spiller, MD FRCP, Study Director — University of Nottingham; Ching Lam, MBChB MRCP, Principal Investigator — University of Nottingham; Klara Garsed, MBChB MRCP, Principal Investigator — University of Nottingham
Locations (1):
- Nottingham Digestive Diseases Centre, University of Nottingham, Nottingham, United Kingdom